CLINICAL TRIAL: NCT05557617
Title: The Role of Periodontitis and Periodontal Bacteria in Development of Dementia
Brief Title: Periodontitis and Periodontal Bacteria in Dementia
Status: Active, not recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 274963
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Dementia; Periodontitis
MeSH Terms: conditions — Alzheimer Disease; Dementia; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid saved at biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Memory clinic cohort: A cohort of 120 individuals that has been investigated for cognitive impairment at the Memory Clinic, Department of Geriatric Medicine, Örebro University Hospital and from which a sample of cerebrospinal fluid has been stored in biobank.

SUMMARY:
The study is designed to inquire whether the presence of periodontitis and different periodontopathogenic bacterial strains are associated with dementia diagnosis and with the degree of cognitive impairment in participants evaluated at a Memory clinic (Minnesmottagning). Specifically, by analyzing cerebrospinal fluid, the investigators intend to clarify whether the alleged mechanisms for Porphyromonas gingivalis in the aetiology of Alzheimer disease (AD) are supported in a Swedish population and whether they are specific for Porphyromonas gingivalis (as compared to other periodontopathogenic bacteria) and Alzheimer type dementia (as compared to other etiological dementia types), respectively.

DETAILED DESCRIPTION:
Purpose and aims

The study is designed to inquire whether the presence of periodontitis and different periodontopathogenic bacterial strains are associated with dementia diagnosis and with the degree of cognitive impairment in patients evaluated at a Memory clinic (Minnesmottagning). Specifically, by analyzing cerebrospinal fluid (CSF) samples, the investigators intend to clarify whether the alleged mechanisms for Porphyromonas gingivalis (P. gingivalis) in the aetiology of AD are supported in a Swedish population and whether they are specific for P. gingivalis (as compared to other periodontopathogenic bacteria) and Alzheimer type dementia (as compared to other etiological dementia types), respectively.

Research questions

In what proportion of Swedish dementia cases is bacterial DNA from periodontal pathogens, antibodies against periodontal pathogens, gingipain protein from P. gingivalis and gingipain enzyme activity found in CSF? Are these bacteriological findings in the CSF more common or more elevated in individuals that received a diagnosis of dementia, as compared to individuals with a lower level of cognitive dysfunction (e.g. mild cognitive impairment, subjective cognitive impairment, or no diagnosis)? Are measurements of cognitive function, e.g. mini-mental state examination (MMSE) scores, correlated with bacteriological findings in the CSF, including gingipain activity? Is the prevalence of periodontitis higher in participants that received a diagnosis of dementia, as compared to participants with a lower level of cognitive dysfunction? Was the prevalence of periodontitis, 5 - 15 years prior to the diagnostic evaluation, higher in participants that received a diagnosis of dementia, as compared to participants with a lower level of cognitive dysfunction? Are measurements of cognitive function, e.g. mini-mental state examination (MMSE) scores, correlated with periodontitis-related findings? In that case, does the correlation depend on the time interval between the periodontal and the cognitive assessments? Are the above bacteriological findings in the CSF more common or more elevated in participants with severe periodontitis, as compared to participants with mild or no periodontitis? Are periodontitis-related findings correlated with bacteriological findings in the CSF, including gingipain activity? In that case, does the correlation depend on the time interval between the periodontal assessments and the CSF sample? Are P. gingivalis-related findings more common or more pronounced than findings related to other periodontal pathogens in any of these potential relationships? Are P. gingivalis-related findings and other bacteriological findings in the CSF more common or more elevated in participants with AD, as compared to participants with non-Alzheimer dementias? Are P. gingivalis-related findings and other bacteriological findings in the CSF correlated with AD-markers in the CSF, such as β-amyloid, tau and phospho-tau?

Participants

The study is based on a cohort of participants that has been investigated for assumed cognitive impairment at the Memory Clinic (Minnesmottagningen), Department of Geriatric Medicine, Örebro University Hospital. The clinical examination includes cognitive tests, brain imaging, etc. A diagnosis of dementia or mild cognitive impairment may be given, but other cases will not receive any of these diagnoses. As a part of these investigations, a lumbar puncture is usually performed to analyze AD-markers in the cerebrospinal fluid (CSF). Approximately 200 lumbar punctures are performed annually, and an aliquot of each sample (1 - 2 mL) is routinely stored in a biobank for 5 years or longer. To the investigators knowledge, at least 300 samples are stored. A retrospective analysis of these CSF samples will form the basis for the investigators biochemical investigations. From these approximately 300 cases we will select 120 participants to include in our study. Those that received a diagnosis of dementia will be the case group, those that did not fulfil dementia criteria (around 25 %) will serve as a control group. Participants with the most complete available clinical data until we reach 120 inclusions will be included.

Data collection

Cognitive function and existing CSF data

The medical records from Minnesmottagningen include results from cognitive tests, e.g. MMSE, Clock Drawing Test, Trail Making Tests, etc. These will be retrieved and registered.

The diagnoses given at Minnesmottagningen, i.e. dementia (if available, also the etiological type of dementia), minor cognitive impairment, other or no diagnosis, will be documented.

The documented results of CSF-analyses of AD-markers, such as β-amyloid, tau and phospho-tau will be retrieved and registered.

Risk factors for Alzheimer disease and periodontitis

From the participants' medical records, information on known risk factors for AD and periodontitis will be collected, notably hypertension, hyperlipidemia, diabetes mellitus, smoking, alcohol consumption, overweight and obesity, coronary heart disease.

Periodontal evaluation

Dental records, including radiographs from the participants' dentists up to 15 years back will be searched for and reviewed. Periodontal status will be assessed by research dentists based on radiographs and clinical examinations extracted from the study participants' dental records.

CSF analyses

These analyses are viewed as explorative. Therefore, the investigators plan interim evaluations after the first 30 results (for each analysis), to estimate the feasibility of continued analysis. Some of the analyses will be performed at laboratories available to the research group, other analyses will be sent to established research laboratories. Analyses will include:

Bacterial DNA from selected species by Polymerase Chain Reaction (PCR). Gingipain analyses with Enzyme-Linked Immunosorbent Assay (ELISA) and with a specific sensor.

Antibodies against selected bacteria with ELISA. Cytokines, chemokines and growth factors with ELISA / Multiplex. The study is planned to include e.g Aggregatibacter actinomycetemcomitans, Tannerella forsythia and Treponema denticola, however, focusing on P. gingivalis.

Statistical considerations

The power analysis is based on a study from 2019. In CSF from 10 individuals with AD, P. gingivalis DNA was detected in seven, but no control CSFs were included. However, in their post-mortem brain parenchyma analyses, P. gingivalis toxins were present in 91-96 % of AD brains and 39-52 % of control brains. The investigators may envisage 70 % positive CSF findings in dementia participants versus 30 % in controls based on this. For 80 % statistical power and α set at 0.05, the investigators would need a minimum sample size of 61 patients. Due to the explorative nature of the investigators study and a number of uncertainties concerning these calculations, the investigators want to include 120 patients in the study, with an interim evaluation of the CSF analyses after 30 analyses.

Statistical analyzes will be carried out in the computer program Statistical Package for the Social Sciences (SPSS) and will include established standard analyzes, e.g. T-tests, Mann-Whitney tests, Pearson and Spearman correlations, logistic and multivariate regressions.

Significance and scientific novelty

The results from this study could provide support for the theory that periodontitis and specific bacteria, implicated in the development of periodontitis, are involved in the pathogenesis and development of dementia. Clarifying the disease mechanisms of Alzheimer's disease and other types of dementia is an important step toward finding more efficient strategies to prevent and treat these diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

- Any person that has been investigated for possible cognitive impairment at Minnesmottagningen, Department of Geriatric Medicine, Örebro University Hospital, and has a CSF sample stored in the biobank. This includes patients who received a diagnosis of dementia (major cognitive disorder) and patients not so diagnosed.

Exclusion Criteria:

* No CSF sample available in biobank
* Incomplete or unavailable clinical and radiological data in medical and dental records, concerning e.g. cognitive tests and AD-biomarker analyses
* Dementia with known etiological diagnosis, e.g. dementia due to alcohol use disorder or traumatic brain injury.
* Creutzfeldt-Jakob disease or other transmissible prion disease
* Non-consenting persons

Ages: 25 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 120 patients that has been investigated for cognitive impairment at the Memory Clinic, Department of Geriatric Medicine, Örebro University Hospital and from which a sample of cerebrospinal fluid has been stored in biobank.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacteriological findings in relation to neurocognitive outcome | 2022-10-01 - 2023-12-31
  The presence of DNA, antibodies and toxins from selected bacterial species in biobank stored cerebrospinal fluid.
Periodontitis in relation to neurocognitive outcome | 2022-10-01 - 2023-12-31
  Retrospectively collected clinical and radiographic periodontal status

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bejerot, Professor, Study Director — Region Örebro County
Locations (1):
- Region Örebro county, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominy SS, Lynch C, Ermini F, Benedyk M, Marczyk A, Konradi A, Nguyen M, Haditsch U, Raha D, Griffin C, Holsinger LJ, Arastu-Kapur S, Kaba S, Lee A, Ryder MI, Potempa B, Mydel P, Hellvard A, Adamowicz K, Hasturk H, Walker GD, Reynolds EC, Faull RLM, Curtis MA, Dragunow M, Potempa J. Porphyromonas gingivalis in Alzheimer's disease brains: Evidence for disease causation and treatment with small-molecule inhibitors. Sci Adv. 2019 Jan 23;5(1):eaau3333. doi: 10.1126/sciadv.aau3333. eCollection 2019 Jan. PMID 30746447